CLINICAL TRIAL: NCT02710305
Title: Randomized Clinical Trial of Oral Hyoscine Butyl Bromide With Cervical Lidocaine Cream in Reducing Pain During Hysterosalpingography
Brief Title: Oral Hyoscine Butyl Bromide With Cervical Lidocaine Cream in Reducing Pain During Hysterosalpingography
Acronym: HBTB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HS1
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Pain Relief

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): oral hyoscine butyl bromide tablets plus lidocaine cream
  Interventions: Drug: oral hyoscine butyl bromide tablets plus lidocaine cream
- Group B (Placebo Comparator): oral placebo tablets plus placebo cream
  Interventions: Drug: oral placebo tablets plus placebo cream

INTERVENTIONS:
Drug: oral hyoscine butyl bromide tablets plus lidocaine cream — patients will take oral hyoscine butyl bromide 30 minutes before the procedure plus lidocaine anesthetic cream placed into their cervix immediately before the procedure
  Arms: Group A
Drug: oral placebo tablets plus placebo cream — patients will take oral placebo 30 minutes before the procedure plus placebo cream placed into their cervix immediately before the procedure
  Arms: Group B

SUMMARY:
hysterosalpingography is a diagnosis procedure in the evaluation of infertile women and considered to be the traditional and the gold standard in the assessment of the patency of the fallopian tubes. The major disadvantage of hysterosalpingography is pain. In a study reported the patients complained of moderate to severe pain during the procedure. It is reported that some patients undergoing hysterosalpingography was more stressful and anxiety and effect on pain scores.

ELIGIBILITY:
Inclusion Criteria:

• The infertile women who indicated for HSG

Exclusion Criteria:

* contraindications to Hyoscine or lidocaine
* known sensitivity to contrast media
* abnormal uterine bleeding
* genital tract infection
* suspected pregnancy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean pain score during HSG | intraoperative

SECONDARY OUTCOMES:
Mean pain score after HSG | 30 minutes
rate of side effects | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided